CLINICAL TRIAL: NCT06932445
Title: Impact of Malnutrition on Liver and Spleen Stiffness in Children Evaluated by Shear Wave Elastography
Brief Title: Effect of Malnutrition on Liver and Spleen Stiffness in Children
Acronym: SWE
Status: Recruiting | Type: Observational
Sponsor: Mehmet Akif AĞIR (Other)
Responsible Party: Sponsor-Investigator, Mehmet Akif AĞIR, Specialist in Pediatric Gastroenterology, Selcuk University
Organization: Selcuk University (Other)
Other Study IDs: 2025/201
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Malnutrition in Children; Liver Stiffness; Spleen Stiffness; Shear Wave Elastography
Keywords: Malnutrition; Liver Stiffness; Spleen Stiffness; Shear Wave Elastography; Children
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malnutrition Group: Children diagnosed with malnutrition based on World Health Organization (WHO) criteria. Participants in this group will undergo shear wave elastography to evaluate liver and spleen stiffness.
  Interventions: Diagnostic Test: Shear Wave Elastography
- Healthy Control Group: Age- and sex-matched healthy children with no known chronic diseases. These participants will also undergo shear wave elastography to allow comparison of organ stiffness values with the malnutrition group.
  Interventions: Diagnostic Test: Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Shear Wave Elastography — Shear wave elastography will be used to measure liver and spleen stiffness in all participants. The procedure will be performed using standard ultrasound-based elastography protocols by a pediatric radiologist.
  Other Names: SWE

SUMMARY:
This prospective observational study aims to evaluate the effect of malnutrition on liver and spleen stiffness in children using shear wave elastography. Two groups of participants will be enrolled: children diagnosed with malnutrition and age-matched healthy controls. Organ stiffness measurements will be compared between the two groups to assess the impact of malnutrition on liver and spleen tissue properties.

DETAILED DESCRIPTION:
This is a prospective observational study designed to investigate the effect of malnutrition on liver and spleen stiffness in children. The study will include two groups: children diagnosed with malnutrition according to WHO criteria, and age- and sex-matched healthy controls without any known chronic illness.

All participants will undergo shear wave elastography (SWE) to measure liver and spleen stiffness using standardized ultrasound protocols. Measurements will be performed by a pediatric radiologist blinded to the nutritional status of the participants.

The primary objective is to compare organ stiffness values between malnourished children and healthy controls. Secondary analyses will explore correlations between severity of malnutrition and stiffness values. The study aims to provide non-invasive insights into early organ-level changes associated with pediatric malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 18 years.
* Diagnosis of malnutrition based on World Health Organization (WHO) criteria (for malnutrition group).
* Healthy children without any chronic illness (for control group).

Exclusion Criteria:

* Children with chronic diseases (e.g., liver disease, diabetes, immunocompromised conditions).
* Children who have previously undergone liver or spleen surgery.
* Children with inability to cooperate during elastography measurement.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will include children aged 6 to 18 years, divided into two groups:
  1. Malnutrition group: Children diagnosed with malnutrition according to World Health Organization (WHO) criteria.
  2. Healthy control group: Age- and sex-matched healthy children with no known chronic illnesses.
  Both groups will undergo shear wave elastography to measure liver and spleen stiffness.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Liver stiffness value (kPa) | At baseline (single time point assessment)
  Liver stiffness will be measured in kilopascals (kPa) using shear wave elastography. The average of three valid measurements will be recorded for each participant.
Spleen stiffness value (kPa) | At baseline
  Spleen stiffness will be measured in kilopascals (kPa) using shear wave elastography. Similar to liver, the average of three valid measurements will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared upon request with qualified researchers, subject to institutional review and approval. Data sharing will be conducted in accordance with the university's data protection policies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2026-January 2028
Access Criteria: The individual participant data (IPD) will be accessible to qualified researchers upon request. Access will be granted following the approval of the Institutional Review Board (IRB) or relevant ethics committee. Researchers will be provided with access to de-identified data, including liver and spleen stiffness measurements, to ensure participant privacy. Access will be granted through a secure data-sharing platform or through direct data transfer from the research team. Data access will be subject to the terms and conditions of the institution's data-sharing policy.